CLINICAL TRIAL: NCT04532346
Title: Safety and Efficacy of Hydroxychloroquine in Children's Interstitial Lung Diseases With Genetic Causes: a Randomized Controlled Study
Brief Title: Hydroxychloroquine in Children's Interstitial Lung Diseases With Genetic Causes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLL202008
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Lung Disease; Surfactant Dysfunction
MeSH Terms: conditions — Lung Diseases, Interstitial; Surfactant Dysfunction | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine in a dose of 10 mg/kg*d, p.o., bid for 12 months. The maximum daily dose is 400mg.
  Interventions: Drug: Hydroxychloroquine
- control (No Intervention): control group which do not take hydroxychloroquine for treatment.

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine Sulfate is an anti-malarial and anti-rheumatic drug. hydroxychloroquine has been reported to improve the clinical status of chILD cases wtih genetic causes. The exact mechanism of action of hydroxychloroquine is unknown. In additon to having anti-inflammatory properties, hydroxychloroquine has been shown to affect intracellular processing of surfactant protein.
  Arms: Hydroxychloroquine

SUMMARY:
The aim of this proposed study is to evaluate the efficacy and safety of hydroxychloroquine (HCQ) in children's interstitial lung diseases(chILD) with genetic causes. This study is a randomized controlled clinical trial.

DETAILED DESCRIPTION:
Children Interstitial lung disease (chILD) is a heterogeneous group of rare respiratory disorders of known and unknown etiologies that are mostly chronic and associated with high morbidity and mortality. Genetic factors are important contributors to chILD. Genetic variations have been mainly described in genes encoding (or interacting with) the surfactant proteins (SP): SP-C (SFTPC) and the ATP-binding cassette-family A-member 3 (ABCA3) (ABCA3), and less frequently in the genes encoding NKX homeobox 2 (NKX2)-1 (NKX2-1), SP-B (SFTPB), SP-A (SFTPA) and other genes.

Hydroxychloroquine has been reported to be useful in cases or case series of chILD including those with genetic causes alone or in combination with systemic steroids. However, the efficacy is highly variable and no randomized controlled study has been reported. The study is a randomized controlled investigation aiming to evaluate the efficacy and safety of hydroxychloroquine in chILD with genetic causes.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of chILD with age<18 years
* Genetically diagnosed (e.g. SFTPC, SFTPB, ABCA3, NKX2-1, CSF2RA, CSF2RB, IARS, MARS, COPA, SLC7A7, LRBA)
* Patients have to be clinically stable with no major changes in their medication in the last 4 weeks
* No HCQ treatment in the last 12 weeks
* Signed and dated informed consent of the subject (if subject has the ability) and the representatives (of underaged children) must be available before start of any specific trial procedures

Exclusion Criteria:

* Acute severe infectious exacerbations
* Known hypersensitivity to HCQ, or other ingredients of the tablets
* Proven retinopathy or maculopathy
* Renal insufficiency at screening, defined as glomerular filtration rate (GFR)< 40 mL/min/1.73 m2 in patients aged 3 to 8 weeks< 60 mL/min/1.73 m2 in patients ≥ 8 weeks of age
* Participation in other clinical trials during the present clinical trial

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Oxygenation status | at first month, at 3rd month, at 6th month, at 12th month
  It is a repeated measurement variable. It is a binary variable (1/0). In a patient without supplemental O2, increase≥5% in O2 saturation or decrease in respiratory rate≥20% means significant change or responder to hydroxychloroquine and the varibale would be setted into "1". In a patient with supplemental O2, increase≥5% in O2 saturation or decrease in respiratory rate≥20% or withdrawal of O2 means significant change or responder to hydroxychloroquine and the varibale would be setted into "1". If no supplemental O2 is necessary, the O2 saturation and respiratory rate are measured in an awake patient after 5 min at rest. If the patient needs supplement O2 , the supplementation is withdrawn after 5 min at rest and the O2 saturation and respiratory rate are measured.

SECONDARY OUTCOMES:
Improvement in clinical manifestation | at first month, at 3rd month, at 6th month, at 12th month
  It is a repeated measurement variable. It is a binary variable (1/0). If coughing resolved, intercostal retraction disappeared and weight for height back to normal is observed in a patient or improvement in chest radiography and pulmonary function tests is present, it means improvement in clinical manifestation and the variable would be setted into "1".

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Kurland G, Deterding RR, Hagood JS, Young LR, Brody AS, Castile RG, Dell S, Fan LL, Hamvas A, Hilman BC, Langston C, Nogee LM, Redding GJ; American Thoracic Society Committee on Childhood Interstitial Lung Disease (chILD) and the chILD Research Network. An official American Thoracic Society clinical practice guideline: classification, evaluation, and management of childhood interstitial lung disease in infancy. Am J Respir Crit Care Med. 2013 Aug 1;188(3):376-94. doi: 10.1164/rccm.201305-0923ST. PMID 23905526
- [Result] Bush A, Cunningham S, de Blic J, Barbato A, Clement A, Epaud R, Hengst M, Kiper N, Nicholson AG, Wetzke M, Snijders D, Schwerk N, Griese M; chILD-EU Collaboration. European protocols for the diagnosis and initial treatment of interstitial lung disease in children. Thorax. 2015 Nov;70(11):1078-84. doi: 10.1136/thoraxjnl-2015-207349. Epub 2015 Jul 1. PMID 26135832
- [Result] Deutsch GH, Young LR, Deterding RR, Fan LL, Dell SD, Bean JA, Brody AS, Nogee LM, Trapnell BC, Langston C; Pathology Cooperative Group; Albright EA, Askin FB, Baker P, Chou PM, Cool CM, Coventry SC, Cutz E, Davis MM, Dishop MK, Galambos C, Patterson K, Travis WD, Wert SE, White FV; ChILD Research Co-operative. Diffuse lung disease in young children: application of a novel classification scheme. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1120-8. doi: 10.1164/rccm.200703-393OC. Epub 2007 Sep 20. PMID 17885266
- [Result] Litao MK, Hayes D Jr, Chiwane S, Nogee LM, Kurland G, Guglani L. A novel surfactant protein C gene mutation associated with progressive respiratory failure in infancy. Pediatr Pulmonol. 2017 Jan;52(1):57-68. doi: 10.1002/ppul.23493. Epub 2016 Jun 30. PMID 27362365
- [Result] Nattes E, Lejeune S, Carsin A, Borie R, Gibertini I, Balinotti J, Nathan N, Marchand-Adam S, Thumerelle C, Fauroux B, Bosdure E, Houdouin V, Delestrain C, Louha M, Couderc R, De Becdelievre A, Fanen P, Funalot B, Crestani B, Deschildre A, Dubus JC, Epaud R. Heterogeneity of lung disease associated with NK2 homeobox 1 mutations. Respir Med. 2017 Aug;129:16-23. doi: 10.1016/j.rmed.2017.05.014. Epub 2017 May 26. PMID 28732825
- [Result] Sun Y, Hu G, Luo J, Fang D, Yu Y, Wang X, Chen J, Qiu W. Mutations in methionyl-tRNA synthetase gene in a Chinese family with interstitial lung and liver disease, postnatal growth failure and anemia. J Hum Genet. 2017 Jun;62(6):647-651. doi: 10.1038/jhg.2017.10. Epub 2017 Feb 2. PMID 28148924
- [Result] Braun S, Ferner M, Kronfeld K, Griese M. Hydroxychloroquine in children with interstitial (diffuse parenchymal) lung diseases. Pediatr Pulmonol. 2015 Apr;50(4):410-9. doi: 10.1002/ppul.23133. Epub 2014 Dec 9. PMID 25491573
- [Result] Kroner C, Reu S, Teusch V, Schams A, Grimmelt AC, Barker M, Brand J, Gappa M, Kitz R, Kramer BW, Lange L, Lau S, Pfannenstiel C, Proesmans M, Seidenberg J, Sismanlar T, Aslan AT, Werner C, Zielen S, Zarbock R, Brasch F, Lohse P, Griese M. Genotype alone does not predict the clinical course of SFTPC deficiency in paediatric patients. Eur Respir J. 2015 Jul;46(1):197-206. doi: 10.1183/09031936.00129414. Epub 2015 Feb 5. PMID 25657025